CLINICAL TRIAL: NCT02775253
Title: Chronic Cold Acclimation Stimulates the Browning of Subcutaneous White Adipose in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiang Guang-da (Other)
Responsible Party: Sponsor-Investigator, Xiang Guang-da, Director of Endocrinol Dept., Wuhan General Hospital of Guangzhou Military Command
Organization: Wuhan General Hospital of Guangzhou Military Command (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016Wze005
Record Dates: First submitted 2016-05-08; First posted 2016-05-17 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Type 2 Diabetes; Cold Acclimation
Keywords: Brown adipose tissue; Subcutaneous white adipose tissue; White adipose tissue
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chronic cold acclimation group (Experimental): All patients will be conducted a chronic cold acclimation intervention for 33 days.
  Interventions: Other: Chronic cold acclimation

INTERVENTIONS:
Other: Chronic cold acclimation

SUMMARY:
Adipose tissues, which include white adipose tissue (WAT) and brown adipose tissue (BAT), play an essential role in regulating whole-body energy homeostasis. Recent studies also reveal the presence of a subset of cells in WAT that could be induced by environmental or hormonal factors to become "brown-like" cells, and this "beigeing" process has been suggested to have strong antiobesity an antidiabetic benefits. More recently, one study showed that Short-term cold acclimation (10 days) improved insulin sensitivity, but did not activate the browning of subcutaneous white adipose in patients with type 2 diabetes mellitus. Here, investigators hypothesize that a chronic cold acclimation can activate the the browning of subcutaneous white adipose in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
All subjects must receive metformin therapy, Patients have chronic cold acclimation intervention for 33 days. During the subsequent cold acclimation period, subjects are exposed to an environmental temperature of 14-15 °C for 33 consecutive days, with cold exposure for 2 h on the first day, 4 h on the second day and 6 h on the third through the 33th day.Biopsy for subcutaneous white adipose and skeletal muscle was performed before and after the intervention program under local anesthesia. The brown fat characteristics and insulin signaling of biopsy samples will be measured. The expression levels of uncoupling protein-1 (UCP-1), peroxisome proliferator-activated receptor r coactivator 1 a (PGC1a), growth factor receptor binding protein-10 (Grb10), PR domain containing 16 (PRDM16) will be determined before and after the intervention programme from the biopsy samples. In addition, a combination of positron emission tomography (PET) and computed tomography (CT) - with the glucose analogue 18F-fluorodeoxyglucose (18F-FDG) as a tracer will be performed for brown adipose tissue before and after the intervention programme.Insulin sensitivity will be checked before and after the intervention programme by insulin clamp assay, and endothelial function will be measured by ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* 18-60 years old
* Body mass index 18.5-28 kg/m2
* HbA1c < 6.5%
* Well controlled diabetes

Exclusion Criteria:

* Type 1 diabetes
* Body mass index < 18.5 kg/m2
* Body mass index > 28 kg/m2
* Female
* Taking any drugs other than metformin
* haemoglobinA1c >=6.50%

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
The changes of UCP-1 expression in subcutaneous white adipose before and after cold acclimation program | From baseline to 33 days
  The expression differences (fold) will be compared before and after cold acclimation program in UCP-1.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan General Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No